CLINICAL TRIAL: NCT05075226
Title: Outcomes of Vivity EDOF IOL Implantation in Patients With Well Controlled OAG or OHT
Brief Title: Visual Outcomes of Vivity in Patients With Well Controlled Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Dr. Paul Harasymowycz, MD, Associate Professor, Maisonneuve-Rosemont Hospital
Other Study IDs: EDOF in POAG
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Vivity Extended Depth of Focus — Cataract surgery

SUMMARY:
Glaucoma is a progressive optic neuropathy that results in a loss of contrast sensitivity and visual field if not detected and treated. When glaucoma patients undergo cataract surgery, they are often not ideal candidates for many existing presbyopia correcting IOLs as they reduce contrast sensitivity because of the splitting of light and are more likely to have visual disturbances secondary to diffractive steps in the IOL design. This is largely because of a higher rate of ocular surface disease and meibomian gland dysfunction in this patient population due to the chronic utilization of topical drops. As a result of this, patients with glaucoma currently receive aspheric monofocal IOLs during cataract surgery, which are lenses with minimal loss of contrast sensitivity but only one point of focus (typically targeted for distance). This necessitates the use of glasses for near and intermediate vision and has an impact on quality of life for these patients.

The Vivity Extended Depth of Focus (EDOF) IOL is a new technology that maintains uncompromised distance vision and provides improved intermediate vision correction, reducing the need for glasses. This lens uses a new optical system with no diffractive steps in the IOL; trials in non-glaucomatous patients have shown the rate of visual aberrations to be comparable to an aspheric monofocal IOL which are currently the standard of care in patients with glaucoma. There is no published data on outcomes of this IOL in patients with primary open angle glaucoma (POAG) or ocular hypertension (OHT). Studies are required to evaluate the clinical success of this new lens technology in glaucomatous patients. This will be the first study in Canada to report clinical outcomes of the Vivity IOL in this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Patients undergoing uncomplicated cataract surgery with IOL implantation
* Patients with both eyes that calculate for IOL powers in the following ranges: 15-25D spherical power (for Vivity)
* Patients possessing with-the-rule or against-the-rule astigmatism ≤2.50 D
* Well controlled OAG or OHT defined as IOP less than or equal to 18mmHg
* Mild to moderate glaucoma as defined by MD VF loss less than 12 dB and no VF defect within the central 5 degrees with 0dB or less than 15dB of both hemi-fields in the central 5 degrees

Exclusion Criteria:

* Ocular comorbidity that might hamper post-operative visual acuity (ie. Macular degeneration, macular edema, uveitis, corneal dystrophy, diabetic retinopathy)
* Ocular trauma or zonula instability
* Previous refractive surgery
* Irregular corneal astigmatism and keratoconus
* Difficulties comprehending written or spoken English or French language
* Patients with physical or intellectual disability
* Patients unable to fixate
* Patients with uncontrolled glaucoma or advanced glaucoma
* Patients that are undergoing filtration or tube surgery or MIGS devices for glaucoma
* Patients with previous filtration or tube surgery for glaucoma
* Patients with unreliable biometry
* Severe dry eye disease or ocular surface disease
* Patients where Barrett Toric Calculator recommends T5 or higher toric IOL

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Prospective, single surgeon, single site (Clinique Bellevue, Montreal)
  * Sample size: Single arm (n=30) 30 bilateral patients (60 eyes total)
  * Patients who underwent bilateral cataract surgery with implantation of Vivity non-toric IOL (15-25D IOL spherical power)
  * Binocular VA endpoints were evaluated at baseline and 3 months postop
  * Visual disturbances (QUVID) and spectacle independence (IOLSAT) questionnaires to be administered at 3 months postop after implantation of second eye
  * Barrett Universal II and Barrett Toric IOL Calculator (for determining exclusion if T3 or higher is calculated) were used for IOL calculation and targeted for emmetropia bilaterally for both groups
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Binocular uncorrected visual acuity | 3 months
  Binocular uncorrected visual acuities at 6m distance will be measured
Binocular uncorrected visual acuity | 3 months
  Binocular uncorrected visual acuities at intermediate distance (66cm) will be measured
Binocular uncorrected visual acuity | 3 months
  Binocular uncorrected visual acuities at near distance (40cm) will be measured

SECONDARY OUTCOMES:
Severity, frequency of bothersomeness of starbursts, haloes, and glare | 3 months
  Severity, frequency of bothersomeness of starbursts, haloes, and glare will be evaluated using the QUVID questionnaire
Spectacle independence | 3 months
  Spectacle independence will be evaluated using the IOLSAT questionnaire
IOP | 1 day
  IOP will be measured in mmHg
IOP | 1 month
  IOP will be measured in mmHg
IOP (mmHg at 1 day, 1 month and 3 months) | 3 months
  IOP will be measured in mmHg
Mean refractive outcomes | 3 months
  Mean refractive outcomes (error and MRSE) will be evaluated
Refractive target accuracy | Approximate patient follow-up time is 4 months following phacoemulsification and insertion of the study lens in the second eye. Time in between eyes will be approximately 1-2 months.
  Percentage of eyes with an APE of 0.50D or less
Contrast sensitivity | pre-operation
  Contrast sensitivity will be evaluated using the Pelli-Robson Chart
Contrast sensitivity | 1 month
  Contrast sensitivity will be evaluated using the Pelli-Robson Chart
Contrast sensitivity | 3 months
  Contrast sensitivity will be evaluated using the Pelli-Robson Chart

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harasymowycz, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Clinique Bellevue, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The plan is to publish the study in an Ophthalmology journal and present the data at national and international ophthalmological conferences (ASCRS 2021/2022, AAO 2021/2022, COS 2022, CGS 2022)